CLINICAL TRIAL: NCT06895863
Title: The Copenhagen Magnetic Personalized Accelerated Brain Circuit Therapy (CoMPACT) Trial
Brief Title: COpenhagen Magnetic Personalized Accelerated Brain Circuit Therapy for Treatment Resistant Depression
Acronym: CoMPACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Research Centre for Magnetic Resonance (Other)
Collaborators: Glostrup University Hospital, Copenhagen (Other); Mental Health Center North Zealand (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CoMPACT; 10.46540/3166-00150B (Other Grant/Funding Number: The Independent Research Fond Denmark); Precision-BCT - 9068-00025A (Other Grant/Funding Number: Innovation Fund Denmark)
Record Dates: First submitted 2025-01-16; First posted 2025-03-26 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Treatment Resistant Depression
Keywords: Brain circuit therapy; Major depressive disorder (MDD); Transcranial magnetic stimulation (TMS); Intermittent theta burst stimulation (iTBS); Copenhagen Magnetic Personalized Accelerated Brain Circuit Therapy (COMPACT); Treatment resistant depression (TRD)
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Double-blinded randomized sham controlled
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Real intermittent theta burst stimulatio (iTBS) of the dorsolateral prefrontal cortex (DLPFC) (Active Comparator)
  Interventions: Device: MagVenture XP Orange Stimulator and active side of MagVenture COOL-B65 coil.
- Real intermittent theta burst stimulation (iTBS) of the left inferior parietal lobule (IPL) (Active Comparator)
  Interventions: Device: Device: MagVenture XP Orange Stimulator and active side of MagVenture COOL-B65 coil.
- Sham Comparator: Sham stimulation to either left IPL (50%) or left DLPFC (50%) (Sham Comparator)
  Interventions: Device: Sham stimulation of the MagVenture MagPro XP Orange Edition Prototype flipping the active side of the MagVenture Cool-B65 coil

INTERVENTIONS:
Device: MagVenture XP Orange Stimulator and active side of MagVenture COOL-B65 coil. — Intermittent theta burst stimulation (iTBS) targeting the left dorsolateral prefrontal cortex (DLPFC) will be administered over five consecutive days.
  On each intervention day, patients will undergo five high frequency iTBS sessions (each lasting approximately 10 minutes, excluding preparation) with about 50 minutes of rest between sessions. Each iTBS session delivers 1,800 pulses, resulting in a total of 25 sessions and 45,000 pulses over the course of a standard work week.
  Arms: Real intermittent theta burst stimulatio (iTBS) of the dorsolateral prefrontal cortex (DLPFC)
Device: Device: MagVenture XP Orange Stimulator and active side of MagVenture COOL-B65 coil. — Intermittent theta burst stimulation (iTBS) targeting the left inferior parietal lobule (IPL) will be administered over five consecutive days using the stimulation pattern described in the active DLPFC arm.
  Arms: Real intermittent theta burst stimulation (iTBS) of the left inferior parietal lobule (IPL)
Device: Sham stimulation of the MagVenture MagPro XP Orange Edition Prototype flipping the active side of the MagVenture Cool-B65 coil — Device: Sham stimulation of the left DLPFC or IPL will be administered using the same stimulation duration and repetition as the active iTBS.
  To match the subjective experience of iTBS, the sham CoMPACT uses a dedicated (Active/Placebo) stimulation coil that has both active and sham functions, generating the same sound level regardless of the type of stimulation.
  Arms: Sham Comparator: Sham stimulation to either left IPL (50%) or left DLPFC (50%)

SUMMARY:
The CoMPACT trial is a randomized double-blinded sham-controlled study aimed at testing a novel accelerated and personalized transcranial Magnetic Stimulation (TMS) treatment for patients with Treatment Resistant Depression (TRD).

CoMPACT consists of 25 sessions of intermittent theta-burst transcranial stimulation (iTBS) consisting of high inter-pulse frequency administered five times daily over five consecutive days.

The trial will include 78 patients with TRD who will be randomly assigned to one of three groups:

* Group 1: Real CoMPACT targeting the left dorsolateral prefrontal cortex (DLPFC).
* Group 2: Real CoMPACT targeting a novel site, the left inferior parietal lobule (IPL).
* Group 3: Sham CoMPACT targeting the left DLPFC (50%, Group 3a) or left IPL (50%, Group 3b).

The hypothesis is that real prefrontal or parietal CoMPACT targeting will significantly alleviate depression symptoms compared to sham targeting, without compromising safety, feasibility, or tolerability.

The trial incorporates a personalized approach, using electrical field (E-field) modeling based on individual structural brain scans to tailor and standardize iTBS, ensuring accurate targeting of cortical volume and consistent induced electrical field strength. To delineate the treatment mechanism of action at the brain network level, multi brain mapping models will be implemented. Electroencephalography (EEG) records of spontaneous and TMS-evoked electrical brain activity will be obtained before, during, and after iTBS sessions to understand how the high frequency burst protocol functionally engages the stimulated cortex. Structural and functional brain MRI before and after the treatment will be used to study changes in depression-related brain networks. This will offer key insights into how CoMPACT affects depression-related brain networks and may identify neuroimaging markers for predicting treatment response, and thus informing future TBS treatments for TRD.

DETAILED DESCRIPTION:
Repetitive TMS (rTMS) of left DLPFC was approved by the US Food and Drug Administration (FDA) in 2008 as a therapy TRD, and this was extended to the equally effective iTBS protocol in 2018.

Dysfunctional connectivity between the left DLPFC and subgenual anterior cingulate cortex (sgACC) has been implicated in the pathogenesis of depression. It has been hypothesized that rTMS-induced neuroplasticity in left DLPFC modifies functional connectivity between left DLPFC and sgACC, normalizing the underlying brain circuit dysfunction.

A recent development has been a move towards "accelerated" rTMS protocols with more than one session per day. Recently, two studies reported promising results for the Stanford Accelerated Intelligent Neuromodulation Treatment (SAINT) protocol for TRD.

The aim of the COMPACT trial is to introduce and test a novel accelerated iTBS therapy for TRD that is designed to significantly expand existing work on accelerated iTBS.

The novel CoMPACT protocol utilizes high frequency bursts to produce a strong "acceleration" effect, securing therapeutic efficacy and clinical feasibility.

The COMPACT protocol consists of five iTBS sessions per day (rather than 10 sessions per day as given in the "SAINT" protocol) over five consecutive days to increase feasibility. In addition to accelerated iTBS of left DLPFC, the invetigators will test clinical efficacy of a novel parietal target, the left IPL. The investigators hypothesize that accelerated iTBS of the area in left IPL that shows a strong negative functional connectivity with the sgACC will be also highly effective in treating TRD compared to the accelerated sham protocol.

Anatomically guided personalized targeting and dosing will be based on E-field modeling informed by the individual cortical anatomy revealed by the patient's structural brain MRI.

Patients with TRD are recruited from psychiatric departments in Copenhagen. Information material with contact details for the project will be available in waiting rooms at the outpatient clinics so that potential participants can contact the project themselves. Furthermore, we will recruit by advertising via Trialtree.dk After inclusion, participants will undergo a baseline assessment (T0) that includes evaluating depression severity and several widely used psychiatric rating scales measuring anhedonia, cognitive deficits, and treatment-related adverse effects. A list of the tests included can be found in the "Outcome" section.

Within two weeks after T0, patients will undergo 5 days of active iTBS targeting either the left DLPFC or the left IPL, or a sham intervention on the left DLPFC or IPL, for a total of 25 sessions. During the first and last day of intervention week, EEG will be used recorded before, during and after first and last iTBS sessions. This helps to investigate acute changes in the cortical activity patterns induced by a single iTBS and the cumulative functional effects on cortical activity caused by the CoMPACT protocol.

Moreover, EEG response to a single and multi TMS pulse, so-called transcranial evoked potentials (TEPs), will be measured before and after iTBS session. This will allow us to explore how high-frequency burst iTBS modulates cortical excitation and inhibition in targeted regions and its potential correlation with clinical response. Online EEG monitoring during iTBS will be performed can also be used to document safety and capture brain activity during the periods separating consecutive iTBS trains.

The antidepressive effects of the intervention (Hamilton Depression Rating Scale as primary outcome) will be assessed, within 3 days after the last session. The rest of the clinical tests will be performed within 5 days after end of treatment (T1). The long-term effect on symptom of depression and other clinical effect will be tested after 4 weeks (T2) and at potential 6 months follow-up.

Assessments at T0 and T1 will also include structural (T1 and T2 weighted sequences), diffusion sensitive MRI, resting-state, and task-based functional MRI (fMRI). Task-related fMRI will reveal how the active CoMPACT intervention modifies brain activity and connectivity within key brain networks compared to sham COMPACT. Cognitive performance will be also probed using a selected set of cognitive tests at T0, T1 and T2.Referral to standard TMS therapy for non-responders:

If patients have not entered remission (i.e. a score less than 7 on HDS-17) immediately after the end of COMPACT treatment or at visit T1, they will be offered standard TMS treatment. A treatment that is approved for general clinical use in psychiatric wards and elsewhere.

Data will be collected at the participating sites in the Capital Region of Denmark (RegionH). After end of trial and final data analysis, anonymized trial-related data and methods will be made available to other researchers through public databases after publication of the main clinical outcome paper in accordance with Danish law.

ELIGIBILITY:
Inclusion criteria:

* Age range between 18 and 95 years
* In- or outpatients with a moderate to severe single episode or periodic MDD according to ICD-10, verified by a M.I.N.I. interview.
* Major Depression Inventory (self-rapport) score higher than 25.
* Lacking or insufficient effect of at least two drug trials from two distinct classes, e.g., SSRI, SNRI, TCA, or MAO-inhibitors, used in the current episode, with adequate dose and duration as judged by the investigator.
* Duration of the current episode must be longer than 2 months but shorter than 4 years, as judged by the investigator.

Exclusion criteria:

* History of neurologic disease affecting the brain, including dementia and epilepsy
* Schizophrenia or any other psychotic disorder except for psychotic depression
* Head trauma causing more than 5 minutes loss of consciousness
* Suicidal or psychotic symptoms making the transport of participants hazardous
* Any form of compulsory admission or treatment within the past three months
* Treatment with ECT in the current depressive episode
* Non-responders to TBS treatment within the current episode
* Current harmful use or dependency of substances according to ICD-10 and interfering with outcome evaluation as judged by investigator's discretion.
* High risk of non-adherence as judged by investigators discretion
* Medical and psychiatric conditions interfering with study outcome and safety as judged by investigator's discretion.
* Female participants of childbearing age must not be pregnant or breast feeding, and they must use contraception during the trial.
* One of the prime contra-indications for MRI, including severe claustrophobia (see Appendix 08.05)
* One of the prime contra-indications for TMS and persons with electrically, magnetically, or mechanically activated implants or with metal or magnetic pieces in their head (see Appendix 08.04)
* Patients who do not wish to be informed about MRI or EEG findings, which may have clinical relevance.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in the Hamilton Rating Scale for Depression-6 (HDS-6) Score | 1) Baseline T0: (1 (+1) week before intervention. 2) Before the first iTBS session on the first day of intervention week. 3) A day after end of intervention (+2 days). 4) Follow-up (T2): 4 weeks after end of intervention.
  The HDS-6 total score reflects the severity of depression, ranging from 0 to 24, with higher scores indicating more severe symptoms.
  0-6 = normal, 7-8= mild depression, 9-11 = moderate depression, 12-22 = severe to very severe depression.
  A 3-point change is considered to be clinically significant, which is a very conservative criterion.

SECONDARY OUTCOMES:
Change in the Hamilton Rating Scale for Depression-17 (HDS-17) Score | 1) Baseline T0: (1 (+1) week before intervention. 2) Before the first iTBS session on the first day of intervention week. 3) A day after end of intervention (+2 days) . 4) Follow-up (T2): 4 weeks after end of intervention.
  The HDS-17 score ranges from 0 to 52, with higher scores reflecting greater depression severity.
  0-7: Normal 8-13: Mild depression 14-18: Moderate depression 19-22: Severe depression
  ≥23: Very severe depression
Change in the WHO-5 Well-being Index (WHO-5) score | 1) Baseline T0: (1 (+1) week before intervention. 2) Postintervention (T1): 3 (+/-2 ) days after end of intervention. 3) Follow-up (T2): 4 weeks after end of intervention.
  The World Health Organization Five Well-being Index (WHO-5) score measures overall well-being on a scale of 0 to 100, with higher scores indicating better well-being.
  Score Interpretation:
  0-28: Poor well-being, possible clinical depression 29-50: Low mood or well-being 51-100: Good well-being
Change Snaith-Hamilton Pleasure Scale (SHAPS) score | 1) Baseline T0: (1 (+1) week before intervention. 2) Postintervention (T1): 3 (+/-2 ) days after end of intervention. 3) Follow-up (T2): 4 weeks after end of intervention.
  SHAPS measure anhedonia. The score ranges from 0 to 14, with higher scores reflecting greater levels of anhedonia
Change in Overall Anxiety Severity and Impairment Scale (OASIS) score | 1) Baseline T0: (1 (+1) week before intervention. 2) Postintervention (T1): 3 (+/-2 ) days after end of intervention. 3) Follow-up (T2): 4 weeks after end of intervention.
  OASIS The score is between 0 and 20. Higher scores indicates greater levels of anxiety and impairment.
Visual analogue mood scale (VAMS) | 1) Baseline T0: (1 (+1) week before intervention. 2) On every day of intervention. 3) Postintervention (T1): 3 (+/-2 ) days after end of intervention. 4) Follow-up (T2): 4 weeks after end of intervention.
  Scale rating mood 1-10. Higher score indicate better mood.
Change in functionality Assessment Short Test (FAST) score | 1) Baseline T0: (1 (+1) week before intervention. 2) Postintervention (T1): 3 (+/-2 ) days after end of intervention. 3) Follow-up (T2): 4 weeks after end of intervention.
  FAST FAST assesses functional impairment. The total score range is 0 to 72. Higher scores indicate greater functional impairment.
Change in Pittsburgh Sleep Quality Index (PSQI) score | Baseline T0: (1 (+1) week before intervention., Postintervention (T1): 3 (+/-2 ) days after end of intervention. Follow-up (T2): 4 weeks after end of intervention.
  PSQI assesses sleep quality. The total score ranges from 0 to 21, with higher scores indicating poorer sleep quality.
TMS Sensation Questionnaire (TMSens_Q) | Intervention week: before and after the first and last sessions on both days 1 and 5
  TMSens_Q assesses and quantifies the sensation and discomfort related to transcranial magnetic stimulation.
Screening for Cognitive Impairment in Psychiatry (SCIP) | 1) Baseline T0: (1 (+1) week before intervention. 2) Postintervention (T1): 3 (+/-2 ) days after end of intervention. 3) Follow-up (T2): 4 weeks after end of intervention.
  The SCIP score ranges from 0 to 75, with lower scores indicating greater cognitive deficits.
Cognitive Complaints in Bipolar Disorder Rating Assessment (COBRA) score | 1) Baseline T0: (1 (+1) week before intervention. 2) Postintervention (T1): 3 (+/-2 ) days after end of intervention. 3) Follow-up (T2): 4 weeks after end of intervention.
  COBRA uses a 4-point scale (no difficulty- severe difficulty). The score ia 0 to 36, with higher scores indicating greater cognitive difficulties.
Aarhus Side effect Assessment Questionnaire (ASAQ) | Baseline T0: (1 (+1) week before intervention. Postintervention (T1): 3 (+/-2 ) days after end of intervention. Follow-up (T2) 4 weeks after end of intervention.
  ASAQ uses a 5-point scale (not at all to very much). The score is from 0 to 27. higher scores indicate greater presence of side effects.
Young Mania Rating scale (YMRS) | Intervention week: before the first session on Day 1 and at the end of each intervention day.
  The Young Mania Rating Scale (YMRS) is used to assess the potential risk of transcranial magnetic stimulation (TMS) inducing mania. It ranges from 0 to 60, with higher scores indicating more severe symptoms.
  0-12: No significant mania 13-19: Mild mania 20-25: Moderate mania
  ≥26: Severe mania
The Stroop Color and Word Test (SCWT) | 1) Baseline T0: (1 (+1) week before intervention. 2) Postintervention (T1): 3 (+/-2 ) days after end of intervention. 3) Follow-up (T2): 4 weeks after end of intervention.
  SCWT uses a 4 point scale (no difficulty to severe difficulty). Fewer errors and faster completion indicate better cognitive control and executive functioning.
Trail Making Test A & B (TMT) | 1) Baseline T0: (1 (+1) week before intervention. 2) On the end of day 1 of intervention week. 3) Postintervention (T1): 3 (+/-2 ) days after end of intervention. 4) Follow-up (T2): 4 weeks after end of intervention.
  TMT-A tests the times to connect all number in correct order. TMT-B tests the total time to alternate between numbers and letters. Fewer errors and faster completion indicate better cognitive control and executive functioning.
Grooved Pegboard Test (GPT) | 1) Baseline T0: (1 (+1) week before intervention. 2) On the end of day 1 of intervention week. 3) Postintervention (T1): 3 (+/-2 ) days after end of intervention. 4) Follow-up (T2): 4 weeks after end of intervention.
  Grooved Pegboard Test (GPT). Fewer errors and faster completion indicate better motor skills.
Treatment Expectation Questionnaire (TEX-Q) | Baseline T0: (1 (+1) week before intervention.
  Question about the patient's expectations for the treatment effect.

OTHER OUTCOMES:
Changes in magnetic resonance imaging (MRI) from baseline to postintervention | 1) Baseline T0: (1 (+1) week before intervention. 2) Postintervention (T1): 3 (+/-2 ) days after end of intervention.
  Structural MRI (sMRI) gives high-resolution images of the brain anatomy and allows for accurate calculation of different volumes of the brain regions.
  Diffusion MRI (dMRI) measures the regional diffusion properties of water and provides micro-structural information on the direction of fiber tracts and structural connectivity in relation to our stimulation targets.
  Functional MRI (fMRI) can map the functional connectivity of the brain during resting periods and during performing reward related tasks.
Changes in Resting-State EEG Power Bands | Intervention week: Before and after first and last sessions on both days 1 and 5
  EEG will be used to assess changes in cortical activity power induced by a single iTBS session, as well as the cumulative effects across an intervention day. The analysis will cover the entire frequency spectrum, with a particular focus on the theta and alpha bands. Additionally, alterations in both periodic and aperiodic components of the power spectrum will be studied.
Immediate changes in EEG power spectrum | Intervention week: During the first and last sessions on both days 1 and 5
  EEG will be used to assess acute changes in cortical power spectrum between consecutive burst trains with a particular focus on the theta and alpha band. Additionally, alterations in both periodic and aperiodic components of the power spectrum will be studied.
Changes in EEG-based Connectivity | Intervention week. Before, during and after the first and last sessions both days 1 and 5
  Exploratory analysis of potential alterations in connectivity within the related network during and after a single iTBS session, compared to baseline. In addition to the investigation of a single session, the cumulative effect of multiple sessions will also be explored.
Changes in TEPs ( transcranial evoked potentials) | Intervention week. Before and after first and last sessions on both days 1 and 5
  TEP measurements (EEG response to single and multiple TMS pulses) will be conducted using active and sham TMS protocols. Changes in TEP components (peaks such as N45, P60, and N100) induced by a single intervention session or across multiple sessions will be studied.
Heart rate variability | Intervention week. During first and last sessions on both days 1 and 5
  Electrocardiography (ECG) will measure changes in heart rate variability (HRV), specifically RR interval variability, during an iTBS session. This will serve as a heart-brain coupling index, which reflects target engagement by assessing autonomic nervous system activity in relation to neural activity.
Patient guess regarding treatment | Postintervention (T1): 3 (+/-2 ) days after end of intervention.
  Questionnaire assessing the patient's guess of whether they have received active or sham stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Hartwig Siebner, Professor, Principal Investigator — Danish Researach Centre for Magnetic Resonance; Poul Videbech, Professor, Principal Investigator — Center for Neuropsychiatric Depression Research, Mental health Center Glostrup
Locations (3):
- Denmark (3):
  - Centre of Neuropsychiatric Depression Research, Glostrup Municipality
  - Mental Health Center North Zealand, Hilleroed
  - Danish Research Centre for Magnetic Resonance, Hvidovre

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cole EJ, Phillips AL, Bentzley BS, Stimpson KH, Nejad R, Barmak F, Veerapal C, Khan N, Cherian K, Felber E, Brown R, Choi E, King S, Pankow H, Bishop JH, Azeez A, Coetzee J, Rapier R, Odenwald N, Carreon D, Hawkins J, Chang M, Keller J, Raj K, DeBattista C, Jo B, Espil FM, Schatzberg AF, Sudheimer KD, Williams NR. Stanford Neuromodulation Therapy (SNT): A Double-Blind Randomized Controlled Trial. Am J Psychiatry. 2022 Feb;179(2):132-141. doi: 10.1176/appi.ajp.2021.20101429. Epub 2021 Oct 29. PMID 34711062
- [Background] Cole EJ, Stimpson KH, Bentzley BS, Gulser M, Cherian K, Tischler C, Nejad R, Pankow H, Choi E, Aaron H, Espil FM, Pannu J, Xiao X, Duvio D, Solvason HB, Hawkins J, Guerra A, Jo B, Raj KS, Phillips AL, Barmak F, Bishop JH, Coetzee JP, DeBattista C, Keller J, Schatzberg AF, Sudheimer KD, Williams NR. Stanford Accelerated Intelligent Neuromodulation Therapy for Treatment-Resistant Depression. Am J Psychiatry. 2020 Aug 1;177(8):716-726. doi: 10.1176/appi.ajp.2019.19070720. Epub 2020 Apr 7. PMID 32252538
- [Background] Voigt JD, Leuchter AF, Carpenter LL. Theta burst stimulation for the acute treatment of major depressive disorder: A systematic review and meta-analysis. Transl Psychiatry. 2021 May 28;11(1):330. doi: 10.1038/s41398-021-01441-4. PMID 34050123
- [Background] Kan RLD, Padberg F, Giron CG, Lin TTZ, Zhang BBB, Brunoni AR, Kranz GS. Effects of repetitive transcranial magnetic stimulation of the left dorsolateral prefrontal cortex on symptom domains in neuropsychiatric disorders: a systematic review and cross-diagnostic meta-analysis. Lancet Psychiatry. 2023 Apr;10(4):252-259. doi: 10.1016/S2215-0366(23)00026-3. Epub 2023 Mar 7. PMID 36898403
- [Background] Ressler KJ, Mayberg HS. Targeting abnormal neural circuits in mood and anxiety disorders: from the laboratory to the clinic. Nat Neurosci. 2007 Sep;10(9):1116-24. doi: 10.1038/nn1944. PMID 17726478
- [Background] Fox MD, Buckner RL, White MP, Greicius MD, Pascual-Leone A. Efficacy of transcranial magnetic stimulation targets for depression is related to intrinsic functional connectivity with the subgenual cingulate. Biol Psychiatry. 2012 Oct 1;72(7):595-603. doi: 10.1016/j.biopsych.2012.04.028. Epub 2012 Jun 1. PMID 22658708
- [Background] Cash RFH, Weigand A, Zalesky A, Siddiqi SH, Downar J, Fitzgerald PB, Fox MD. Using Brain Imaging to Improve Spatial Targeting of Transcranial Magnetic Stimulation for Depression. Biol Psychiatry. 2021 Nov 15;90(10):689-700. doi: 10.1016/j.biopsych.2020.05.033. Epub 2020 Jun 7. PMID 32800379